CLINICAL TRIAL: NCT01940523
Title: Randomized Controlled Trial of Tranexamic Acid in Total Knee Arthroplasty: Intravenous vs. Topical
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital for Special Surgery, New York (Other)
Collaborators: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 12166; NCT02123095 (obsolete NCT alias)
Record Dates: First submitted 2013-09-09; First posted 2013-09-12 (Estimated); Results first posted 2017-06-14 (Actual); Last update posted 2019-11-27 (Actual); Status verified 2019-11

CONDITIONS: Osteoarthritis
Keywords: total knee arthroplasty; total knee replacement; tranexamic acid; osteoarthritis; degenerative joint disease
MeSH Terms: conditions — Osteoarthritis; Joint Diseases | interventions — Tranexamic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Topical Tranexamic Acid (Active Comparator): 3 vials of tranexamic acid (1g tranexamic acid in 10cc each) must be mixed in the operating room by the team at the start of surgery with 45cc of saline solution (for a total of 3g tranexamic acid in 75mL solution). This solution will be applied to the open joint surfaces with two 60mL syringes (one with 60mL and one with 15m). The solution will be left in contact with the tissues for five minutes. The surgeon will suction away excess solution. The site may be irrigated before or after the tranexamic acid bath as long as the solution is in contact for at least five full minutes. After that, the tourniquet will be released and the rest of the surgery will proceed according to the standard of care.
  Interventions: Drug: Topical Tranexamic Acid
- Intravenous Tranexamic Acid (Active Comparator): 1 vial (1g of IV tranexamic acid in 10mL solution) will be administered prior to inflation of the tourniquet. A second 1g dose of IV tranexamic acid will be given during initiation of the closure after the tourniquet is deflated and during closure.
  Interventions: Drug: Intravenous Tranexamic Acid

INTERVENTIONS:
Drug: Topical Tranexamic Acid — 3 vials of tranexamic acid (1g tranexamic acid in 10cc each) must be mixed in the operating room by the team at the start of surgery with 45cc of saline solution (for a total of 3g tranexamic acid in 75mL solution). This solution will be applied to the open joint surfaces with two 60mL syringes (one with 60mL and one with 15m). The solution will be left in contact with the tissues for five minutes. The surgeon will suction away excess solution. The site may be irrigated before or after the tranexamic acid bath as long as the solution is in contact for at least five full minutes. After that, the tourniquet will be released and the rest of the surgery will proceed according to the standard of care.
  Arms: Topical Tranexamic Acid
Drug: Intravenous Tranexamic Acid — 1 vial (1g of IV tranexamic acid in 10mL solution) will be administered prior to inflation of the tourniquet. A second 1g dose of IV tranexamic acid will be given during initiation of the closure after the tourniquet is deflated and during closure.
  Arms: Intravenous Tranexamic Acid

SUMMARY:
The purpose of this study is to determine whether topical or intravenous administration of tranexamic acid during unilateral total knee replacement is more effective at reducing bleeding in the first 24 hours following surgery. Tranexamic acid is a synthetic drug that has been shown to reduce blood drain output and the need for blood transfusions in both its topical and intravenous forms and is commonly used in orthopedic surgery. We hypothesize that IV and topical administration of tranexamic acid will be equally good at reducing the loss of blood and the need for transfusion immediately following total knee replacement.

DETAILED DESCRIPTION:
This randomized controlled trial compares the blood loss of patients undergoing unilateral total knee replacements who randomly receive either the topical or the intravenous form of tranexmamic acid during surgery. Patients in the intravenous arm of the study will receive 1 gram of tranexamic acid in 10 milliliters of solution prior to inflation of the tourniquet and 1 gram of tranexamic acid in 10 milliliters of solution during closure. For patients in the topical arm of the study, prior to the release of the tourniquet they will receive 3 grams of tranexamic acid in 75ccs of solution directly on the site of the incision.

The primary result measurement will be blood drain output from the knee at 24 hours after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Primary total knee replacmeent
* Osteoarthritis
* Unilateral

Exclusion Criteria:

* Revision surgery
* Donated preoperative autologous blood
* On chronic anticoagulation medication such as Coumadin, Xarelto, Plavix, or Aspirin (other than 81mg)
* Preoperative hepatic or renal dysfunction
* Diagnosis of inflammatory disease
* Diagnosis of inflammatory arthritis
* Pregnant
* Breastfeeding
* Preoperative hemoglobin <10g/dL
* International Normalized Ratio>1.4
* Abnormal Partial Thromboplastin Time
* Preoperative platelet count of <150,000mm^3
* Creatinine > 1.4

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 640 (Actual)
Dates: Start 2013-05 (Actual); Primary Completion 2015-12-28 (Actual); Study Completion 2017-05-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Mayman, MD, Principal Investigator — Hospital for Special Surgery, New York
Locations (2):
- United States (2):
  - Mayo Clinic, Rochester, Minnesota
  - Hospital for Special Surgery, New York, New York

RESULTS

PARTICIPANT FLOW:
Groups:
- Topical Tranexamic Acid: 3 vials of tranexamic acid (1g tranexamic acid in 10cc each) must be mixed in the operating room by the team at the start of surgery with 45cc of saline solution (for a total of 3g tranexamic acid in 75mL solution). This solution will be applied to the open joint surfaces with two 60mL syringes (one with 60mL and one with 15m). The solution will be left in contact with the tissues for five minutes. The surgeon will suction away excess solution. The site may be irrigated before or after the tranexamic acid bath as long as the solution is in contact for at least five full minutes. Tourniquet will be released.
  Topical Tranexamic Acid: 3 vials of tranexamic acid (1g tranexamic acid in 10cc each) must be mixed in the operating room by the team at the start of surgery with 45cc of saline solution (for a total of 3g tranexamic acid in 75mL solution). This solution will be applied to the open joint surfaces with two 60mL syringes (one with 60mL and one with 15m).
Period: Overall Study
Arm/Group | Topical Tranexamic Acid | Intravenous Tranexamic Acid
Started | 320 | 320
Completed | 320 | 320
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Topical Tranexamic Acid: 3 vials of tranexamic acid (1g tranexamic acid in 10cc each) must be mixed in the operating room by the team at the start of surgery with 45cc of saline solution (for a total of 3g tranexamic acid in 75mL solution). This solution will be applied to the open joint surfaces with two 60mL syringes (one with 60mL and one with 15m).
  Topical Tranexamic Acid: 3 vials of tranexamic acid (1g tranexamic acid in 10cc each) must be mixed in the operating room by the team at the start of surgery with 45cc of saline solution (for a total of 3g tranexamic acid in 75mL solution). This solution will be applied to the open joint surfaces with two 60mL syringes (one with 60mL and one with 15m). The solution will be left in contact with the tissues for five minutes.
- Total: Total of all reporting groups
Arm/Group | Topical Tranexamic Acid | Intravenous Tranexamic Acid | Total
Number analyzed (Participants) | 320 | 320 | 640
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 146 | 151 | 297
  >=65 years | 174 | 169 | 343
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.87 (9.42) | 66.35 (9.16) | 66.6 (9.28)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: The overall enrollment for the study is N=640
  Participants
    Female | 193 | 187 | 380
    Male | 127 | 133 | 260

OUTCOME MEASURES:

1. Primary Outcome: Total Blood Loss
Description: The amount of blood lost during surgery is the primary outcome measure. Blood loss is determineusing an equation that calculates the patient's blood volume based on their height and weight, then multiplies the patient's blood volume by the change in their hematocrit after surgery compared to before surgery.
Time Frame: during surgery
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | Topical Tranexamic Acid | Intravenous Tranexamic Acid
Number analyzed (Participants) | 320 | 320
ml | 323.59 (255.89) | 271.22 (212.06)

2. Secondary Outcome: Drain Output
Description: The amount of blood collected by a drain attached to the knee is measured 24 hours after surgery.
Time Frame: from end of surgery to 24 hours postoperatively
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | Topical Tranexamic Acid | Intravenous Tranexamic Acid
Number analyzed (Participants) | 320 | 320
ml | 560.13 (297.21) | 456.22 (275.39)

3. Secondary Outcome: The Number Patients Requiring a Transfusion
Description: TThe number Patients requiring a transfusion over the course of the patient's hospital stay.
Time Frame: over course of hospital stay (averaging three days)
Measure: Count of Participants; unit: Participants
Groups:
- IV TXA Group; Topical TXA Group: Kaitlin - Explain this group....
Arm/Group | IV TXA Group | Topical TXA Group
Number analyzed (Participants) | 320 | 320
Participants | 2 | 6

ADVERSE EVENTS:
Time Frame: During the hospital stay, adverse event data was collected
Arm/Group | Topical Tranexamic Acid | Intravenous Tranexamic Acid
Serious Adverse Events (participants affected / at risk) | 0/320 | 0/320
Other Adverse Events (participants affected / at risk) | 0/320 | 0/320

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes